CLINICAL TRIAL: NCT05071313
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Study to Evaluate the Immunogenicity and Safety of Ad26.RSV.preF-based Vaccine and High-dose Seasonal Influenza Vaccine, With and Without Coadministration, in Adults Aged 65 Years and Older
Brief Title: A Study of an Ad26.RSV.preF-based Vaccine and High-dose Seasonal Influenza Vaccine, With and Without Coadministration, in Adults Aged 65 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR109064; VAC18193RSV3005 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2021-09-28; First posted 2021-10-08 (Actual); Results first posted 2023-09-13 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Influenza, Human Prevention; Respiratory Syncytial Viruses Prevention
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Coadministration (CoAd) Group (Experimental): Participants will receive Ad26.RSV.preF-based vaccine and quadrivalent high dose influenza vaccine concomitantly on Day 1 and placebo on Day 29.
  Interventions: Biological: Ad26.RSV.preF-based vaccine; Biological: Quadrivalent High-dose Influenza Vaccine; Biological: Placebo
- Group 2: Control Group (Experimental): Participants will receive placebo and quadrivalent high-dose influenza vaccine on Day 1 and Ad26.RSV.preF-based vaccine on Day 29.
  Interventions: Biological: Ad26.RSV.preF-based vaccine; Biological: Quadrivalent High-dose Influenza Vaccine; Biological: Placebo

INTERVENTIONS:
Biological: Ad26.RSV.preF-based vaccine — Ad26.RSV.preF-based vaccine will be administered as single IM injection.
Biological: Quadrivalent High-dose Influenza Vaccine — Quadrivalent High-dose Influenza Vaccine will be administered as IM injection.
Biological: Placebo — Placebo will be administered as IM injection to Ad26.RSV.preF-based vaccine.

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of Ad26.RSV.preF-based vaccine and quadrivalent high-dose seasonal influenza vaccine when administered either concomitantly or separately.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to adhere to the prohibitions and restrictions specified in this protocol
* In the investigator's clinical judgment, the participant must be in stable health at the time of vaccination. Participants will be included on the basis of medical history and vital signs performed between informed consent from (ICF) signature and vaccination
* Before randomization, a participant must be not intending to conceive by any methods, postmenopausal or surgically sterile
* From the time of vaccination through 3 months after vaccination, agrees not to donate blood
* Must be willing to provide verifiable identification, have means to be contacted and to contact the investigator during the study
* Participant must be able to work with smartphones/tablets/computers

Exclusion Criteria:

* History of malignancy within 5 years before screening not in the following categories: a) participants with squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix may be enrolled at the discretion of the investigator; b) participants with a history of malignancy within 5 years before screening, with minimal risk of recurrence per investigator's judgement, can be enrolled
* Known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or their excipients (including specifically the excipients of the study vaccine)
* History of severe allergic reactions (example, anaphylaxis) to any component of the Quadrivalent high-dose influenza vaccine, including egg protein, or following a previous dose of any influenza vaccine
* Has abnormal function of the immune system resulting from either clinical condition, chronic or recurrent use of systemic corticosteroids within 2 months prior to study vaccination, or immunomodulating agents within 6 months prior to study vaccination
* Per medical history, participant has chronic active hepatitis B or hepatitis C infection
* History of acute polyneuropathy (example, Guillain-Barre syndrome) or chronic idiopathic demyelinating polyneuropathy
* Has a serious chronic disorder, example, chronic obstructive pulmonary disease or congestive heart failure, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, Alzheimer's disease, or has any condition, including conditions placing the participant at high risk for severe influenza, for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments
* Received vaccination with seasonal influenza vaccine for the current influenza season in the Northern Hemisphere

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 777 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2022-10-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (19):
- United States (19):
  - Ark Clinical Research, Long Beach, California
  - Research Centers of America, LLC, Hollywood, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Synexus Clinical Research US Inc, The Villages, Florida
  - Synexus Clinical Research US Inc, Chicago, Illinois
  - Meridian Clinical Research, LLC, Rockville, Maryland
  - Sundance Clinical Research, St Louis, Missouri
  - Synexus Clinical Research US Inc, St Louis, Missouri
  - Meridian Clinical Research, LLC, Grand Island, Nebraska
  - Meridian Clinical Research, LLC, Lincoln, Nebraska
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Tekton Research Inc., Yukon, Oklahoma
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - VitaLink Research Spartanburg, Spartanburg, South Carolina
  - AMR New Orleans, Formerly New Orleans Center for Clinical Research - New Orleans, an AMR company, Knoxville, Tennessee
  - Optimal Research, Austin, Texas
  - Tekton Research Inc., Austin, Texas
  - DM Clinical Research, Tomball, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV + Placebo (CoAd Group): Participants received intramuscular (IM) injection containing both adenovirus serotype 26 pre-fusion conformation-stabilized F protein (Ad26.RSV.preF) 1*10^11 viral particles (vp) and respiratory syncytial virus prefusion F-protein (RSV preF protein) 150 micrograms (mcg) coadministered with Fluzone high-dose (HD) quadrivalent (QIV) 240 mcg IM injection on Day 1 (vaccination 1) followed by placebo IM injection on Day 29 (vaccination 2).
- Group 2: Placebo With Fluzone HD QIV + Ad26/Protein preF RSV Vaccine (Control Group): Participants received placebo IM injection coadministered with Fluzone HD QIV 240 mcg IM injection on Day 1 (vaccination 1) followed by an IM injection containing both Ad26.RSV.preF 1*10^11 vp and RSV preF protein 150 mcg on Day 29 (vaccination 2).
Period: Overall Study
Arm/Group | Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV + Placebo (CoAd Group) | Group 2: Placebo With Fluzone HD QIV + Ad26/Protein preF RSV Vaccine (Control Group)
Started | 389 | 388
Received Ad26/Protein preF RSV Vaccine With Fluzone in CoAd Group at Day 1 | 385 | 0
Received Placebo With Fluzone in Control Group at Day 1 | 0 | 386
Received Placebo in CoAd Group at Day 29 | 357 | 0
Received Ad26/Protein preF RSV Vaccine in Control Group at Day 29 | 0 | 363
Completed | 355 | 355
Not Completed | 34 | 33
Not completed — Lost to Follow-up | 17 | 10
Not completed — Physician Decision | 1 | 6
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 10 | 15
Not completed — Other | 1 | 0
Not completed — Randomized but not vaccinated | 4 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who received at least 1 study vaccination, regardless of the occurrence of protocol deviations and vaccine type (seasonal influenza, Ad26/protein preF RSV vaccine, or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV + Placebo (CoAd Group) | Group 2: Placebo With Fluzone HD QIV + Ad26/Protein preF RSV Vaccine (Control Group) | Total
Number analyzed (Participants) | 385 | 386 | 771
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.4 (4.94) | 70.7 (4.72) | 70.5 (4.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 223 | 208 | 431
  Male | 162 | 178 | 340
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 33 | 72
  Not Hispanic or Latino | 339 | 344 | 683
  Unknown or Not Reported | 7 | 9 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 38 | 39 | 77
  White | 336 | 333 | 669
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 3 | 6 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 385 | 386 | 771

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Hemagglutination Inhibition (HI) Antibodies Against Each of the Four Influenza Vaccine Strains as Measured by HI Assay
Description: Hemagglutination is a phenomenon by which the hemagglutinin protein of influenza viruses can bind to sialic acid receptors on the red blood cell membrane, thereby forming clumps and is the basis for the HI assay. GMTs of HI antibodies against each of the four influenza vaccine strains as measured by HI assay at 28 days after the administration of a quadrivalent high-dose seasonal influenza vaccine (fluzone) were reported. The analysis was performed on 2 influenza A strains [A/Victoria and A/Tasmania] and 2 influenza B strains [B/Washington and B/Phuket]).
Time Frame: 28 days after vaccination with Fluzone on Day 1 (Day 29)
Population: Per-protocol influenza immunogenicity (PPII) set included all randomized participants who received the first study vaccination, and for whom immunogenicity data are available for at least one of the influenza strains in the vaccine. Samples taken after participant experienced major protocol deviation expected to impact the immunogenicity outcomes were excluded from this analysis, including those who were collected out of window.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV + Placebo (CoAd Group) | Group 2: Placebo With Fluzone HD QIV + Ad26/Protein preF RSV Vaccine (Control Group)
Number analyzed (Participants) | 338 | 338
Titers
  A/Victoria | 178 [145 to 217] | 179 [146 to 219]
  A/Tasmania | 111 [89 to 139] | 123 [98 to 155]
  B/Washington | 93 [74 to 117] | 84 [67 to 106]
  B/Phuket | 38 [31 to 47] | 37 [30 to 46]
Statistical Analysis 1: Comparison: Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV + Placebo (CoAd Group) vs Group 2: Placebo With Fluzone HD QIV + Ad26/Protein preF RSV Vaccine (Control Group); A/Victoria; Test type: Non-Inferiority — Non-inferiority of Group 2 versus Group 1 in terms of the HI antibody titers against all four influenza vaccine strains 28 days after vaccination with fluzone, using a non-inferiority margin of 1.5 for the GMT ratio (Group 2/Group 1); Geometric Mean Ratio = 1.01, 95% CI 2-sided [0.89 to 1.14]
Statistical Analysis 2: Comparison: Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV + Placebo (CoAd Group) vs Group 2: Placebo With Fluzone HD QIV + Ad26/Protein preF RSV Vaccine (Control Group); A/Tasmania; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 1.11, 95% CI 2-sided [0.97 to 1.28]
Statistical Analysis 3: Comparison: Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV + Placebo (CoAd Group) vs Group 2: Placebo With Fluzone HD QIV + Ad26/Protein preF RSV Vaccine (Control Group); B/Washington; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 0.91, 95% CI 2-sided [0.79 to 1.05]
Statistical Analysis 4: Comparison: Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV + Placebo (CoAd Group) vs Group 2: Placebo With Fluzone HD QIV + Ad26/Protein preF RSV Vaccine (Control Group); B/Phuket; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Geometric Mean Ratio = 0.97, 95% CI [0.85 to 1.10]

2. Primary Outcome: GMTs of Prefusion F-protein (preF) Antibodies as Assessed by Enzyme-linked Immunosorbent Assay (ELISA) on Day 29
Description: GMTs of preF antibodies at 28 days after the administration of Ad26.RSV.preF-based vaccine as assessed by ELISA on Day 29 were reported. This outcome measure was planned to be analyzed for specified arm only.
Time Frame: 28 days after vaccination with Ad26.RSV.preF-based vaccine on Day 1 (Day 29)
Population: Per-protocol RSV immunogenicity (PPRI) set included all randomized participants who received Ad26/protein preF RSV vaccine in combination with seasonal influenza vaccine in the CoAd group and Ad26/protein preF RSV vaccine alone in the control group and for which RSV immunogenicity data were available. Samples taken after participant experienced major protocol deviation expected to impact immunogenicity outcomes were excluded from this analysis, including those who were collected out of window.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per liter (EU/L)
Arm/Group | Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV + Placebo (CoAd Group)
Number analyzed (Participants) | 338
ELISA units per liter (EU/L) | 2665 [2209 to 3216]

3. Primary Outcome: GMTs of PreF Antibodies as Assessed by Enzyme-linked Immunosorbent Assay (ELISA) on Day 57
Description: GMTs of preF antibodies at 28 days after the administration of Ad26.RSV.preF-based vaccine as assessed by ELISA on Day 57 were reported. This outcome measure was planned to be analyzed for specified arm only.
Time Frame: 28 days after vaccination with Ad26.RSV.preF-based vaccine on Day 29 (Day 57)
Population: The PPRI set included all randomized participants who received Ad26/protein preF RSV vaccine in combination with seasonal influenza vaccine for the CoAd group and Ad26/protein preF RSV vaccine alone for the control group and for whom RSV immunogenicity data were available. Samples taken after participant experienced major protocol deviation expected to impact the immunogenicity outcomes were excluded from this analysis, including those who were collected out of window.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/L
Arm/Group | Group 2: Placebo With Fluzone HD QIV + Ad26/Protein preF RSV Vaccine (Control Group)
Number analyzed (Participants) | 318
EU/L | 3206 [2648 to 3881]

4. Secondary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) After Study Vaccination 1
Description: Number of participants with solicited local AEs after study vaccination 1 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, were used to assess the reactogenicity of the study vaccine and were pre-defined local (injection site). Solicited local AEs were reported separately for all vaccines because fluzone and RSV vaccine mixture (containing both Ad26. RSV. preF 1*10^11 vp and RSV preF protein 150 mcg) in group 1 were administered in opposite arms on Day 1. Similarly, fluzone and placebo in group 2 were administered in opposite arms on Day 1. Hence, the data for this outcome measure was analyzed separately for each vaccine.
Time Frame: Up to 7 days after study vaccination 1 on Day 1 (Day 8)
Population: The full analysis set (FAS) included all participants who received at least 1 study vaccination, regardless of the occurrence of protocol deviations and vaccine type (seasonal influenza, Ad26/protein preF RSV vaccine, or placebo). Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Fluzone HD QIV (CoAd Group); Group 2: Fluzone HD QIV (Control Group): Participants received Fluzone HD QIV 240 mcg IM injection on Day 1 on right arm.
- Group 1: Ad26/Protein preF RSV Vaccine (CoAd Group): Participants received IM injection containing both Ad26. RSV. preF 1*10^11 vp and RSV preF protein 150 mcg on Day 1 on left arm.
- Group 2: Placebo (Control Group): Participants received placebo as an IM injection on Day 1 on left arm.
Arm/Group | Group 1: Fluzone HD QIV (CoAd Group) | Group 1: Ad26/Protein preF RSV Vaccine (CoAd Group) | Group 2: Fluzone HD QIV (Control Group) | Group 2: Placebo (Control Group)
Number analyzed (Participants) | 371 | 371 | 373 | 373
Participants | 237 | 263 | 219 | 98

5. Secondary Outcome: Number of Participants With Solicited Local AEs After Study Vaccination 2
Description: Number of participants with solicited local AEs after study vaccination 2 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited local AEs that included injection site pain/tenderness, erythema and swelling at the study vaccine injection site, were used to assess the reactogenicity of the study vaccine and were pre-defined local (injection site).
Time Frame: Up to 7 days after study vaccination 2 on Day 29 (Day 36)
Population: The FAS included all participants who received at least 1 study vaccination, regardless of the occurrence of protocol deviations and vaccine type (seasonal influenza, Ad26/protein preF RSV vaccine, or placebo). Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Placebo (CoAdGroup): Participants received placebo as an IM injection on Day 29.
- Group 2: Ad26/Protein preF RSV Vaccine (Control Group): Participants received IM injection containing both Ad26. RSV. preF 1*10^11 vp and RSV preF protein 150 mcg on Day 29.
Arm/Group | Group 1: Placebo (CoAdGroup) | Group 2: Ad26/Protein preF RSV Vaccine (Control Group)
Number analyzed (Participants) | 341 | 343
Participants | 53 | 241

6. Secondary Outcome: Number of Participants With Solicited Systemic AEs After Study Vaccination 1
Description: Number of participants with solicited systemic AEs after study vaccination 1 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Solicited systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants were specifically questioned and which were noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: Up to 7 days after study vaccination 1 on Day 1 (Day 8)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV (CoAd Group): Group 1: Ad26/protein preF RSV vaccine with Fluzone HD QIV (CoAd Group) Participants received intramuscular (IM) injection containing both Ad26. RSV. preF; 1*10^11 viral particles (vp) and RSV preF protein; 150 micrograms (mcg) coadministered with Fluzone high-dose (HD) quadrivalent (QIV) 240 mcg IM injection on Day 1.
- Group 2: Fluzone HD QIV With Placebo (Control Group): Participants received Fluzone HD QIV 240 mcg IM injection coadministered with placebo IM injection on Day 1.
Arm/Group | Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV (CoAd Group) | Group 2: Fluzone HD QIV With Placebo (Control Group)
Number analyzed (Participants) | 371 | 373
Participants | 285 | 181

7. Secondary Outcome: Number of Participants With Solicited Systemic AEs After Study Vaccination 2
Description: Number of participants with solicited systemic AEs after study vaccination 2 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Systemic events included events such as fatigue, headache, nausea, and myalgia, for which participants will be specifically questioned and which will be noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: Up to 7 days after study vaccination 2 on Day 29 (Day 36)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Groups:
- Group 2: Ad26/Protein preF RSV Vaccine (Control Group): Participants received IM injection containing both Ad26. RSV. preF 1*10^11 viral particles and RSV preF protein; 150 mcg on Day 29.
Arm/Group | Group 1: Placebo (CoAdGroup) | Group 2: Ad26/Protein preF RSV Vaccine (Control Group)
Number analyzed (Participants) | 341 | 343
Participants | 80 | 218

8. Secondary Outcome: Number of Participants With Unsolicited AEs After Study Vaccination 1
Description: Number of participants with unsolicited AEs after study vaccination 1 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant was not specifically questioned in the participant diary.
Time Frame: Up to 28 days after study vaccination 1 on Day 1 (Day 29)
Population: The FAS included all participants who received at least 1 study vaccination, regardless of the occurrence of protocol deviations and vaccine type (seasonal influenza, Ad26/protein preF RSV vaccine, or placebo).
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV (CoAd Group): Participants received IM injection containing both Ad26. RSV. preF; 1*10^11 viral particles and RSV preF protein; 150 mcg coadministered with Fluzone HD QIV 240 mcg IM injection on Day 1.
- Group 2: Fluzone HD QIV With Placebo (Control Group): Participants received Fluzone high-dose (HD) quadrivalent (QIV) 240 micrograms (mcg) intramuscular (IM) injection coadministered with placebo IM injection on Day 1.
Arm/Group | Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV (CoAd Group) | Group 2: Fluzone HD QIV With Placebo (Control Group)
Number analyzed (Participants) | 385 | 386
Participants | 57 | 61

9. Secondary Outcome: Number of Participants With Unsolicited AEs After Study Vaccination 2
Description: Number of participants with unsolicited AEs after study vaccination 2 were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Unsolicited AEs were all AEs for which the participant was not specifically questioned in the participant diary.
Time Frame: Up to 28 days after study vaccination 2 on Day 29 (Day 57)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Placebo (CoAdGroup) | Group 2: Ad26/Protein preF RSV Vaccine (Control Group)
Number analyzed (Participants) | 357 | 363
Participants | 34 | 35

10. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) Up to Study Vaccination 1
Description: Number of participants with SAEs up to study vaccination 1 were reported. SAE is any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: From Day 1 up to Day 29
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV (CoAd Group) | Group 2: Fluzone HD QIV With Placebo (Control Group)
Number analyzed (Participants) | 385 | 386
Participants | 2 | 2

11. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs) Up to Study Vaccination 2
Description: Number of participants with SAEs up to study vaccination 2 were reported. SAE is any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: From Day 29 up to 6 months after study vaccination 2 (up to 7 months)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: Placebo (CoAd Group): Participants received placebo IM injection on Day 29.
Arm/Group | Group 1: Placebo (CoAd Group) | Group 2: Ad26/Protein preF RSV Vaccine (Control Group)
Number analyzed (Participants) | 357 | 363
Participants | 11 | 11

12. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI) Up to Study Vaccination 1
Description: Number of participants with AESI up to study vaccination 1 were reported. Thrombosis with thrombocytopenia syndrome (TTS) was considered to be an AESI.
Time Frame: From Day 1 up to Day 29
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Groups:
- Group 2: Fluzone HD QIV With Placebo (Control Group): Participants received Fluzone HD QIV 240 mcg intramuscular (IM) injection coadministered with placebo IM injection on Day 1.
Arm/Group | Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV (CoAd Group) | Group 2: Fluzone HD QIV With Placebo (Control Group)
Number analyzed (Participants) | 385 | 386
Participants | 0 | 0

13. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI) Up to Study Vaccination 2
Description: Number of participants with AESI up to study vaccination 2 were reported. Thrombosis with thrombocytopenia syndrome (TTS) was considered to be an AESI.
Time Frame: From Day 29 up to 6 months after study vaccination 2 (up to 7 months)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Placebo (CoAd Group) | Group 2: Ad26/Protein preF RSV Vaccine (Control Group)
Number analyzed (Participants) | 357 | 363
Participants | 0 | 0

14. Secondary Outcome: Number of Seroconverted Participants After 28 Days of Administration of Influenza Vaccine
Description: Number of seroconverted participants after 28 days of administration of influenza vaccine (fluzone) were reported. Seroconversion is defined for each of the 4 influenza vaccine strains at 28 days after the administration of a quadrivalent high-dose seasonal influenza vaccine: HI titer greater than or equal to (>=) 1:40 in participants with a pre-vaccination HI titer of less than (<) 1:10, or a >=4-fold HI titer increase in participants with a pre-vaccination HI titer of >=1:10.
Time Frame: 28 days after vaccination with fluzone on Day 1 (up to Day 29)
Population: PPII set included all randomized participants who received the first study vaccination, and for whom immunogenicity data were available for at least one of the influenza strains in the vaccine. Samples taken after participant experienced major protocol deviation expected to impact the immunogenicity outcomes were excluded from this analysis, including those who were collected out of window.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV + Placebo (CoAd Group) | Group 2: Placebo With Fluzone HD QIV + Ad26/Protein preF RSV Vaccine (Control Group)
Number analyzed (Participants) | 338 | 338
Participants
  A/Victoria | 203 | 190
  A/Tasmania | 150 | 165
  B/Washington | 134 | 117
  B/Phuket | 79 | 84

15. Secondary Outcome: Number of Seroprotected Participants After 28 Days of Administration of Influenza Vaccine
Description: Number of seroprotected participants after 28 days of administration of influenza vaccine (fluzone) were reported. Seroprotection is defined for each of the 4 influenza vaccine strains as HI titer >=1:40 at 28 days after the administration of a quadrivalent high-dose seasonal influenza vaccine.
Time Frame: 28 days after vaccination with fluzone on Day 1 (up to Day 29)
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV + Placebo (CoAd Group) | Group 2: Placebo With Fluzone HD QIV + Ad26/Protein preF RSV Vaccine (Control Group)
Number analyzed (Participants) | 338 | 338
Participants
  A/Victoria | 323 | 313
  A/Tasmania | 282 | 285
  B/Washington | 247 | 245
  B/Phuket | 117 | 122

ADVERSE EVENTS:
Time Frame: From Day 1 up to 7 months
Description: The full analysis set (FAS) included all participants who received at least 1 study vaccination, regardless of the occurrence of protocol deviations and vaccine type (seasonal influenza, Ad26/protein preF RSV vaccine, or placebo).
Groups:
- Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV (CoAd Group): Participants received intramuscular (IM) injection containing both Ad26. RSV. preF; 1*10^11 viral particles (vp) and RSV preF protein; 150 micrograms (mcg) coadministered with Fluzone high-dose (HD) quadrivalent (QIV) 240 mcg IM injection on Day 1.
Arm/Group | Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV (CoAd Group) | Group 2: Fluzone HD QIV With Placebo (Control Group) | Group 1: Placebo (CoAd Group) | Group 2: Ad26/Protein preF RSV Vaccine (Control Group)
All-Cause Mortality (participants affected / at risk) | 0/385 | 0/386 | 1/357 | 0/363
Serious Adverse Events (participants affected / at risk) | 2/385 | 2/386 | 11/357 | 11/363
Other Adverse Events (participants affected / at risk) | 18/385 | 12/386 | 1/357 | 10/363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV (CoAd Group) (N=385) | Group 2: Fluzone HD QIV With Placebo (Control Group) (N=386) | Group 1: Placebo (CoAd Group) (N=357) | Group 2: Ad26/Protein preF RSV Vaccine (Control Group) (N=363)
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Jaundice Cholestatic (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Covid-19 (Infections and infestations) | 0 | 0 | 1 | 2
Covid-19 Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis Pneumococcal (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia Staphylococcal (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 4
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lung Carcinoma Cell Type Unspecified Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Brain Injury (Nervous system disorders) | 0 | 0 | 0 | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Ad26/Protein preF RSV Vaccine With Fluzone HD QIV (CoAd Group) (N=385) | Group 2: Fluzone HD QIV With Placebo (Control Group) (N=386) | Group 1: Placebo (CoAd Group) (N=357) | Group 2: Ad26/Protein preF RSV Vaccine (Control Group) (N=363)
Chills (General disorders) | 11 | 4 | 1 | 8
Hypertension (Vascular disorders) | 7 | 8 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/13/NCT05071313/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-05): https://cdn.clinicaltrials.gov/large-docs/13/NCT05071313/SAP_001.pdf